CLINICAL TRIAL: NCT02635542
Title: Prospective, Randomized Trial Comparing Effect of General Anesthesia With and Without Neuromuscular Blockade on Postoperative Pulmonary Complications in Elective Cardiac Surgical Patients
Brief Title: Effect of Neuromuscular Blockade on Pulmonary Complications in Elective Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-1016
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Neuromuscular Blockade; Postoperative Complications
Keywords: Postoperative Pulmonary Complications; Residual Neuromuscular Blockade; Cardiac Surgical Procedures
MeSH Terms: conditions — Postoperative Complications; Delayed Emergence from Anesthesia | interventions — Succinylcholine; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Open label drug administration. Outcomes assessor and care providers are otherwise masked.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group CIS (Active Comparator): Continual neuromuscular blockade (standard therapy) during general anesthesia will be provided with cisatracurium (CIS), with 0.2mg/kg IV given as an initial dose and repeated dosing determined by neuromuscular blockade monitoring (peripheral nerve stimulator maintained at 1-2 twitches).
  Interventions: Drug: Cisatracurium
- Group SUX (Experimental): A single dose of neuromuscular blockade (experimental group) will be provided at the start of anesthesia with succinylcholine (SUX), with 1mg/kg IV given as an initial dose and no repeat dosing.
  Interventions: Drug: Succinylcholine

INTERVENTIONS:
Drug: Succinylcholine — Succinylcholine will be used to facilitate endotracheal intubation for general anesthesia in the operating room. No additional neuromuscular blockade will be provided during general anesthesia.
  Other Names: Suxamethonium
  Arms: Group SUX
Drug: Cisatracurium — Cisatracurium will be used to maintain neuromuscular blockade during general anesthesia.
  Other Names: Nimbex
  Arms: Group CIS

SUMMARY:
The investigators will conduct a prospective, randomized trial to assess the impact of neuromuscular blockade on early (<72 hours post-ICU admission) postoperative respiratory complications in cardiac surgical patients. The study will compare continual neuromuscular blockade with cisatracurium to a single dose of succinylcholine during general anesthesia for cardiac surgery.

DETAILED DESCRIPTION:
Residual neuromuscular blockade during the immediate postoperative period is an important patient safety issue. Although used to facilitate the technical performance of surgery, clinical studies have associated neuromuscular blockade (NMB) with increased incidence of postoperative respiratory complications. This effect is likely mediated by residual neuromuscular blockade interfering with airway tone and respiratory effort, leading to postoperative pneumonia, atelectasis or aspiration. However, the vast majority of these studies have involved non-cardiac patient populations, yet patients undergoing cardiac surgery are even more susceptible to the detrimental effects of residual neuromuscular blockade for a number of reasons. Despite widespread utilization of paralysis during cardiac surgery, very little is known about residual neuromuscular blockade in patients following cardiac surgery. Previously published clinical studies date from over a decade ago or are based on retrospective databases from non-cardiac surgery patients, precluding generalizable conclusions. Given the substantial role of neuromuscular blockade in the traditional management of cardiac surgical patients, prospective data is needed to determine the veracity of this association as well as the surgical tolerability of protocols that minimize intraoperative paralysis. The investigators will conduct a prospective, randomized trial to assess impact of neuromuscular blockade on early (<72 hours post-ICU admission) postoperative respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery (CABG, valve replacement, CABG + valve) requiring cardiopulmonary bypass

Exclusion Criteria:

* Emergency surgery
* Extremes of age
* Previous cardiac surgery
* Clinical contraindications to succinylcholine or cisatracurium
* Anticipated difficult tracheal intubation
* Preoperative mechanical ventilation
* Preoperative pharmacologic/mechanical hemodynamic support

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Gerlach, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group CIS | Group SUX
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group CIS | Group SUX | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (14.5) | 64.1 (14.6) | 65.1 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 36 | 29 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Euroscore [Mean (Standard Deviation); unit: units on a scale] — The additive Euroscore (European System for Cardiac Operative Risk Evaluation) is a measure of predicted operative mortality for patients undergoing cardiac surgery. The score is comprised of patient-related factors, cardiac-related factors, and operation-related factors. Higher scores indicate greater risk for operative mortality (possible range 0-43).
  units on a scale | 5.56 (3.08) | 5.28 (3.08) | 5.42 (3.07)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.2 (6.9) | 28.2 (5.9) | 29.2 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Pulmonary Complications
Description: Having at least one of the following complications, determined according to pre-specified criteria: extubation delayed >24hrs, reintubation, mechanical respiratory support, pneumonia, aspiration, ARDS (Acute Respiratory Distress Syndrome), or mortality from respiratory arrest.
Time Frame: 72 hours following surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group CIS | Group SUX
Number analyzed (Participants) | 50 | 50
Participants | 8 | 8
Statistical Analysis 1: Comparison: Group CIS vs Group SUX; Test type: Superiority; p = 1.00, Chi-squared

2. Secondary Outcome: Surgical Conditions
Description: Assessed by surgeon questionnaire designed for study to determine any negative effects impeding the progress of surgery or safety, on scale of 1=poor to 5=excellent
Time Frame: During general anesthesia
Population: 2 participants in the CIS group and 4 participants in the SUX group had missing data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group CIS | Group SUX
Number analyzed (Participants) | 48 | 46
units on a scale | 4.96 (0.20) | 4.65 (0.85)
Statistical Analysis 1: Comparison: Group CIS vs Group SUX; Test type: Superiority; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Group CIS | Group SUX
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02635542/Prot_SAP_000.pdf